CLINICAL TRIAL: NCT02119468
Title: Phase I/II Trial of MLN9708 Plus Pomalidomide and Dexamethasone for Relapsed or Relapsed Refractory Multiple Myeloma
Brief Title: Ixazomib Plus Pomalidomide and Dexamethasone in Treating Patients With Relapsed or Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12267; NCI-2014-00803 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12267 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Refractory Plasma Cell Myeloma; Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Dexamethasone; Calcium Dobesilate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (3mg MLN9708) (Experimental): Patients receive 3mg ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixazomib citrate; Drug: dexamethasone; Drug: pomalidomide
- Treatment (4mg MLN9708) (Experimental): Patients receive 4mg ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixazomib citrate; Drug: dexamethasone; Drug: pomalidomide

INTERVENTIONS:
Drug: ixazomib citrate — Given orally
  Other Names: MLN9708; proteasome inhibitor MLN9708
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: pomalidomide — Given orally
  Other Names: CC-4047; Pomalyst

SUMMARY:
This phase I/II trial studies the side effects and best dose of ixazomib and to see how well it works when given together with pomalidomide and dexamethasone in treating patients with relapsed or relapsed/refractory multiple myeloma. Ixazomib may stop the growth of cancer by interfering with proteasomes (the protein breakdown mechanism in the cells). Pomalidomide and dexamethasone can modify and regulate the immune system and may stop cancer cells from growing. Giving ixazomib with pomalidomide and dexamethasone may be an effective treatment for relapsed or relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) of MLN9708 (ixazomib), when given in combination with pomalidomide and dexamethasone, in patients with relapsed or relapsed/refractory multiple myeloma. (Phase I) II. To estimate the response rate and to evaluate the antitumor activity of the three drug combination: MLN9708 (at the RP2D), pomalidomide and dexamethasone, in patients with relapsed or relapsed/refractory multiple myeloma. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety of MLN9708 at each dose level when given as part of a three drug combination by assessing the following: type, frequency, severity, attribution, time course and duration of adverse events; and clinical laboratory tests at various points in the study. (Phase I) II. To characterize and evaluate toxicities, including type, frequency, severity, attribution, time course and duration, at the RP2D, for the three drug combination. (Phase II) III. To obtain estimates of response duration, depth of response, clinical benefit response, and survival (overall and progression-free), at the RP2D, for the three drug combination. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of ixazomib followed by a phase II study.

Patients receive ixazomib orally (PO) on days 1, 8, and 15; dexamethasone PO on days 1, 8, 15, and 22; and pomalidomide PO on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting pomalidomide or MLN9708 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide or MLN9708 through 90 days after the last dose of study drug; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 90 days after the last dose of study drug; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* All patients enrolled into this trial, must be registered in and must comply with all requirements of the POMALYST (pomalidomide) Risk Evaluation and Mitigation Strategy (REMS) program
* Patients must have a diagnosis of relapsed or relapsed and refractory multiple myeloma with a minimum of one prior regimen and a maximum of 5 prior regimens
* Patients must have had therapy with a proteasome inhibitor and lenalidomide and be refractory to lenalidomide according to the International Myeloma Working Group (IMWG) criteria definition of refractory disease (progressive disease on or within 60 days of stopping lenalidomide)
* Patients must have measurable disease defined as one of the following:

  * Serum M protein >= 0.5 g/dL
  * Urine M protein >= 200 mg/24 hours
  * Serum free light chain >= 10 mg/dL provided the free light chain (FLC) ratio is abnormal
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 75,000/uL for patients in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count >= 50,000/uL for patients in whom >= 50% of bone marrow nucleated cells are plasma cells; platelet transfusions are not allowed within 3 days of last platelet assessment to confirm eligibility
* Total bilirubin =< 1.5 × the institutional upper limit of the normal range (IULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 × IULN
* Calculated creatinine clearance >= 45 mL/min

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (ie, =< grade 1 toxicity) from the reversible effects of prior chemotherapy
* Prior therapy with a combination regimen containing pomalidomide except the 2 drug combination of pomalidomide and dexamethasone
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708
* Central nervous system involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Unable or unwilling to undergo antithrombotic prophylaxis
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 or pomalidomide including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy with evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has > grade 2 peripheral neuropathy on clinical examination during the screening period
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial (for all other standard therapies, no treatment within 14 days of the start of this trial)
* Patients who are pomalidomide refractory, defined as patients who progress on or within 60 days of pomalidomide when given as a single agent or with dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Krishnan, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level #1 (3mg MLN9708): Patients receive ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ixazomib citrate: Given orally
  dexamethasone: Given orally
  pomalidomide: Given orally
- Dose Level #2 (4mg MLN9708): Patients receive ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level #1 (3mg MLN9708) | Dose Level #2 (4mg MLN9708)
Started | 7 | 25
Completed | 7 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level #2 (4mg MLN9708): Patients receive ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ixazomib citrate: Given orally
  dexamethasone: Given orally
  pomalidomide: Given orally
- Total: Total of all reporting groups
Arm/Group | Dose Level #1 (3mg MLN9708) | Dose Level #2 (4mg MLN9708) | Total
Number analyzed (Participants) | 7 | 25 | 32
Age, Continuous [Median (Full Range); unit: years] | 53 [48 to 74] | 63 [38 to 84] | 62 [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 5 | 15 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 23 | 29
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 7 | 20 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 25 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-Limiting Toxicities (Phase I)
Description: Dose Limiting Toxicity (DLT) is defined as any of the toxicities in Section 7.3 that are at least possibly related to either Pomalidomide or MLN9708 that occur during cycle 1. Toxicity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.03. The highest dose level that produces 1/6 dose-limiting toxicities (DLTs) in course 1 will be the maximum tolerated dose (MTD). The RP2D of ixazomib and pomalidomide will generally be the MTD, but it may be less than the MTD based on a review of available data/cumulative toxicities from phase I.
Time Frame: From the initial treatment to Day 28 (Cycle #1)
Population: Patients were considered evaluable for DLT if receiving at least 75% of both Pomalidomide and MLN9708 and followed for the full 28 days during cycle 1 or experience a DLT. All patients who are not evaluable for DLT were replaced.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level #1: 3mg MLN9708; Dose Level #2: 4mg MLN9708: Patients receive ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level #1: 3mg MLN9708 | Dose Level #2: 4mg MLN9708
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

2. Primary Outcome: Overall Response Rate at the Recommended Phase II Dose (RP2D)
Description: Over response rate is calculated as the percent of evaluable patients that have confirmed stringent complete remission (sCR), complete remission (CR), very good partial remission (VGPR) or partial remission [PR]) per modified IMWG criteria. sCR as defined below plus normal FLC ratio and absence of clonal cells in bone marrow. CR defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. VGPR defined as serum and urine M-protein detectable or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h. PR defined as > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h. The exact 95% confidence intervals are calculated for the estimate.
Time Frame: From the initial treatment to 24 months
Population: Patients received 4 mg MLN9708, 4mg pomalidomide, and 40 mg dexamethasone (RP2D).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Groups:
- Dose Level #2 (4mg MLN9708): Patients receive 4mg ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level #2 (4mg MLN9708)
Number analyzed (Participants) | 25
Percentage of Participants (%) | 48 [27.8 to 68.7]

3. Primary Outcome: Maximum Tolerated Dose (MTD) of MLN9708 (Phase I)
Description: The highest dose level that produces 1/6 dose-limiting toxicities (DLTs) in Cycle #1 will be the maximum tolerated dose (MTD). The RP2D of ixazomib and pomalidomide will generally be the MTD, but it may be less than the MTD based on a review of available data/cumulative toxicities from phase I.
Time Frame: From the initial treatment to Day 28 (Cycle #1)
Population: 6 patients treated at dose level #2 in Phase I are evaluable for dose limiting toxicity.
Measure: Number; unit: mg
Arm/Group | Dose Level #2 (4mg MLN9708)
Number analyzed (Participants) | 6
mg | 4

4. Secondary Outcome: Duration of Response at the Recommended Phase II Dose (RP2D)
Description: Time from the date of first documented response (sCR/CR/VGPR or PR) to documented disease relapse, progression or death whichever occurs first. sCR as defined below plus normal FLC ratio and absence of clonal cells in bone marrow. CR defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. VGPR defined as serum and urine M-protein detectable or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h. PR defined as > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h.
Time Frame: Time interval from the date of first documented response (sCR/CR/VGPR or PR) to documented disease relapse, progression or death whichever occurs first, up to 24 months
Population: Patients received 4 mg MLN9708, 4mg pomalidomide, and 40 mg dexamethasone (RP2D).
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Level #2 (4mg MLN9708)
Number analyzed (Participants) | 25
Months | 9.2 [0.9 to 13.9]

5. Secondary Outcome: Clinical Benefit Response Rate at the Recommended Phase II Dose (RP2D)
Description: Clinical benefit response rate is calculated as the percent of evaluable patients that have confirmed stringent complete remission (sCR), complete remission (CR), very good partial remission (VGPR), partial remission (PR), minimal response (MR) or stable disease (SD) per modified IMWG criteria. The exact 95% confidence intervals are calculated for the estimate.
Time Frame: From the initial treatment up to 24 months
Population: Patients received 4 mg MLN9708, 4mg pomalidomide, and 40 mg dexamethasone (RP2D).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Dose Level #2 (4mg MLN9708)
Number analyzed (Participants) | 25
Percentage of Participants (%) | 76 [54.9 to 90.6]

6. Secondary Outcome: One-Year Overall Survival at the Recommended Phase II Dose (RP2D)
Description: Overall survival (OS) was measured from initial treatment to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula.
Time Frame: Date of first dose of study drug to date of death from any cause, up to 24 months. And the median follow-up for the surviving patients is at least one year.
Population: Patients received 4 mg MLN9708, 4mg pomalidomide, and 40 mg dexamethasone (RP2D).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Dose Level #2 (4mg MLN9708)
Number analyzed (Participants) | 25
Percentage of Participants (%) | 82 [59 to 93]

7. Secondary Outcome: One-Year Progression-Free Survival at the Recommend Phase II Dose (RP2D)
Description: Progression-free survival (PFS) was defined as time from initial treatment to recurrence, progression or death. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works. Progression-free survival was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula [Breslow NE, Day NE. Statistical methods in cancer research: volume II, the design and analysis of cohort studies. IARC Sci Publ 1987;82:1-406.]
Time Frame: Date of first dose of study drug to first documented disease relapse, progression or death from any cause, whichever occurs first, up to 24 months. And the median follow-up for the surviving patients is at least one year.
Population: Patients received 4 mg MLN9708, 4mg pomalidomide, and 40 mg dexamethasone (RP2D).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Dose Level #2 (4mg MLN9708)
Number analyzed (Participants) | 25
Percentage of Participants (%) | 34 [16 to 53]

ADVERSE EVENTS:
Time Frame: From the date of the first dose up to 2 years
Groups:
- Dose Level #1 (3mg MLN9708): Patients receive 3mg ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ixazomib citrate: Given orally
  dexamethasone: Given orally
  pomalidomide: Given orally
- Dose Level #2 (4mg MLN9708): Patients receive 4mg ixazomib citrate (MLN9708) orally on days 1, 8, and 15; dexamethasone orally on days 1, 8, 15, and 22; and pomalidomide orally on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ixazomib citrate: Given orally
  dexamethasone: Given orally
  pomalidomide: Given orally
Arm/Group | Dose Level #1 (3mg MLN9708) | Dose Level #2 (4mg MLN9708)
All-Cause Mortality (participants affected / at risk) | 4/7 | 6/25
Serious Adverse Events (participants affected / at risk) | 4/7 | 11/25
Other Adverse Events (participants affected / at risk) | 7/7 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level #1 (3mg MLN9708) (N=7) | Dose Level #2 (4mg MLN9708) (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level #1 (3mg MLN9708) (N=7) | Dose Level #2 (4mg MLN9708) (N=25)
Anemia (Blood and lymphatic system disorders) | 6 (17) | 19 (88)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (8) | 1 (4)
Sinus tachycardia (Cardiac disorders) | 2 (5) | 2 (2)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (2) | 5 (24)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (11)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (13)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 10 (35)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 9 (20)
Dry mouth (Gastrointestinal disorders) | 2 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 4 (8)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (8) | 10 (26)
Vomiting (Gastrointestinal disorders) | 2 (4) | 5 (9)
Chills (General disorders) | 2 (3) | 3 (3)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (3) | 6 (22)
Fatigue (General disorders) | 5 (10) | 15 (79)
Fever (General disorders) | 3 (6) | 3 (6)
Flu like symptoms (General disorders) | 2 (4) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 1 (1) | 3 (4)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 3 (5)
Lung infection (Infections and infestations) | 1 (2) | 2 (2)
Nail infection (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (2) | 7 (12)
Bruising (Injury, poisoning and procedural complications) | 1 (4) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (7)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (8) | 1 (17)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (12) | 1 (4)
Blood bilirubin increased (Investigations) | 3 (5) | 4 (13)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 4 (11) | 4 (21)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (20) | 1 (2)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 6 (24) | 13 (46)
Neutrophil count decreased (Investigations) | 5 (39) | 17 (105)
Platelet count decreased (Investigations) | 5 (43) | 19 (95)
Weight gain (Investigations) | 2 (22) | 2 (10)
Weight loss (Investigations) | 0 (0) | 2 (3)
White blood cell decreased (Investigations) | 6 (40) | 16 (83)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (5) | 11 (20)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 5 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (11) | 6 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (13) | 2 (9)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 4 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (10) | 5 (21)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (20) | 3 (13)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 8 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 6 (34)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (29)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (7) | 7 (12)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 2 (15)
Dizziness (Nervous system disorders) | 3 (5) | 8 (15)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (3) | 5 (6)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (4)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (20) | 12 (59)
Somnolence (Nervous system disorders) | 1 (1) | 1 (7)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 1 (12) | 2 (17)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (7)
Confusion (Psychiatric disorders) | 0 (0) | 5 (36)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (12) | 5 (17)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (5) | 2 (6)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (50) | 5 (37)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 6 (45)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (16)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (122) | 7 (42)
Hypotension (Vascular disorders) | 0 (0) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT02119468/Prot_SAP_000.pdf